CLINICAL TRIAL: NCT06140979
Title: Efficacy of Visual Focusing Game on Children With Attention Deficit Hyperactivity Disorder and Mechanisms of Functional Near-Infrared Spectroscopic Imaging
Brief Title: Visual Focused Play Intervention for Children With ADHD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KY20232300-F-1
Record Dates: First submitted 2023-11-12; First posted 2023-11-21 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Intervention Model Description: The patients in the test group will be given a visual focus game to play and the patients in the control group will be given an animated video of the game that had no therapeutic effect.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Group (Experimental): The patients in the test group will be given a visual focus game to play, and the treatment will be required at least 5 times per week for 2 weeks, with each session lasting 30 minutes.
  Interventions: Behavioral: Playing the game
- Control Group (Sham Comparator): The patients in the control group were given an animated video of the game that had no therapeutic effect, and the video will be required at least 5 times per week for 2 weeks, with each session lasting 30 minutes.
  Interventions: Behavioral: Watching the gameplay video

INTERVENTIONS:
Behavioral: Playing the game — The intervention is based on a parkour game in which the player runs forward as a cartoon character, avoiding obstacles in front of him/her while collecting gold coins and various props. In this process, players need to stay focused and operate in time to avoid obstacles or collect rewards, and as time goes on, the difficulty of the game increases until eventually they cannot avoid obstacles. As time goes on, the difficulty of the game will increase until the end of the game when you can't avoid the obstacles.
  Arms: Test Group
Behavioral: Watching the gameplay video — The intervention consists of a 30-minute non-therapeutic video of a parkour game, which is paused every 10 minutes and requires the patient to click "continue" until the end of the video. No other action is required.
  Arms: Control Group

SUMMARY:
This is a single-center, randomized, double-blind, sham-controlled study that will recruit children with attention deficit hyperactivity disorder and randomly assign them to a test group and a control group. The patients in the test group will be given a visual focus game to play and the patients in the control group will be given an animated video of the game that had no therapeutic effect. Treatment will be required at least 5 times per week for 2 weeks, with each game or video session lasting 30 minutes. Clinical scales and functional near-infrared spectroscopic imaging will be performed before and at the end of the 2 weeks of treatment, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Meeting the diagnostic criteria for ADHD in the U.S. Diagnostic and Statistical Manual of Mental Disorders, 5th edition (DSM-5);
* Aged 6-14 years old;
* Right-handedness (habitual or good use of the right hand in daily life, work, study and labor activities);
* Voluntarily agree to sign an informed consent form;

Exclusion Criteria:

* Wechsler Intelligence Scale for Children (WISC) <80 points;
* The cranial CT or MRI found that there are clear infarction foci, soft foci, occupations and other organic lesions;
* Suffering from serious physical diseases or other severe mental diseases, such as schizophrenia, bipolar disorder, etc;
* Inability to cooperate with fNIRS data collection

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2023-11-10 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in Attention Deficit Hyperactivity Disorder Rating Scale scores between baseline and post-treatment | Baseline and 2 weeks
  The Attention Deficit Hyperactivity Disorder Rating Scale is commonly used to determine whether children have symptoms of ADHD, how severe they are, and how impaired they are. As such, it is a combination of symptom and functional impairment ratings (e.g., unless it is at least moderately impaired to rate a 2 or 3 on a symptom). This is usually done by the clinician based on information provided by the parent/guardian or teacher.

SECONDARY OUTCOMES:
Change in the Parent Symptom Questionnaire scores between baseline and post-treatment | Baseline and 2 weeks
  The Parent Symptom Questionnaire is a child behavior rating scale for parents developed by Conners that is easy to understand and takes parents only 5 to 10 minutes to complete. The scale is primarily used to assess attention deficit hyperactivity disorder in children and can reflect the effectiveness of treatment.
Changes in Functional Near-Infrared Spectral Imaging between Baseline and Post-Treatment | Baseline and 2 weeks
  Functional near-infrared spectroscopic imaging is a safe and fast screening method. It reflects brain activity by measuring blood oxygen levels in the cerebral cortex with promptness, accuracy, and short duration.

CONTACTS AND LOCATIONS:
Overall Officials: Min Cai, Principal Investigator — The First Affiliated Hospital of the Air Force Medical University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Anguera JA, Boccanfuso J, Rintoul JL, Al-Hashimi O, Faraji F, Janowich J, Kong E, Larraburo Y, Rolle C, Johnston E, Gazzaley A. Video game training enhances cognitive control in older adults. Nature. 2013 Sep 5;501(7465):97-101. doi: 10.1038/nature12486. PMID 24005416
- [Result] Barkley RA. Attention-deficit/hyperactivity disorder, self-regulation, and time: toward a more comprehensive theory. J Dev Behav Pediatr. 1997 Aug;18(4):271-9. PMID 9276836
- [Result] Pandian GSB, Jain A, Raza Q, Sahu KK. Digital health interventions (DHI) for the treatment of attention deficit hyperactivity disorder (ADHD) in children - a comparative review of literature among various treatment and DHI. Psychiatry Res. 2021 Mar;297:113742. doi: 10.1016/j.psychres.2021.113742. Epub 2021 Jan 19. PMID 33515870
- [Result] Kollins SH, Childress A, Heusser AC, Lutz J. Effectiveness of a digital therapeutic as adjunct to treatment with medication in pediatric ADHD. NPJ Digit Med. 2021 Mar 26;4(1):58. doi: 10.1038/s41746-021-00429-0. PMID 33772095